CLINICAL TRIAL: NCT03629639
Title: Metformin for Treatment of Psoriasis Combined With Disorders of Glucose and Lipid Metabolism: A Double-Blind, Randomized, Placebo-Controlled Study
Brief Title: Metformin for Treatment of Psoriasis Combined With Disorders of Glucose and Lipid Metabolism
Acronym: MPGLM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-MET/CSU/PSO
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis Vulgaris With Metabolic Disorders
Keywords: Psoriasis; Metformin; Gut microbiota
MeSH Terms: conditions — Psoriasis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): the distributed subjects will be orally administered Metformin 500mg bid lasting for 12 weeks.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): the distributed subjects will be orally administered Metformin-like placebo 500mg bid lasting for 12 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — An intervention of either metformin or placebo 500mg twice daily plus standard care for 12 weeks. Besides Metformin, standardized topical treatment is given to all patients; For severe psoriasis patients(PASI>8), Methotrexate will be treated orally 7.5mg every week for both the intervention group and the placebo group as a systemic standard care.

SUMMARY:
Psoriasis and metabolic disorders are well-known mutual comorbidities. The investigators hypothesized metformin can ameliorate both psoriasis and metabolic disorders mainly via gut microbiota modulation. The investigators design a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of treatment of metformin for psoriasis combined with disorders of glucose and lipid metabolism and to explore the role of gut microbiota during the process.

ELIGIBILITY:
Inclusion Criteria:

criteria 1 and 2 are both needed for inclusion:

1. included if all of the following criteria are met

   * ≥18 years and ≤75 years
   * Diagnosed according to Classification criteria for Psoriasis Vulgaris
   * Understanding the whole process of the study, voluntary participation and signed the informed consent
2. included if at least one of the following criteria is met

   * Body Mass Index (BMI) over 24
   * impaired glucose or insulin resistance

Exclusion Criteria:

* Pregnant women, or women who ready for pregnancy or lactating;
* Have special primary endocrine system lesions that can influence glucose or lipid metabolism
* More than 20% change of their predrug body weight within a half year
* Severe diabetes which needs combined therapy
* Known major systemic diseases like cancer, liver or kidney malfunction, etc.
* Alcohol abuse
* Known severe or chronic infections like tuberculosis or HIV
* Use of other systemic medication that could influence the metabolic level
* Patients participated in any clinical trials within 3 months
* Other cases which researchers believe that can not enroll

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving a Greater Than or Equal to 75 Percentage Improvement From Baseline in Psoriasis Area and Severity Index (PASI 75) Score at Week 12 [ Time Frame: Baseline and Week 12 ] | baseline, Week 12
  Number of participants achieving greater than or equal to 75 percentage improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12. PASI is the widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) -72 (worst). Baseline visit refers to Week 0.

SECONDARY OUTCOMES:
improvement of dermatology quality of life: Dermatology Life Quality Index | baseline, Week 12
  Evaluated by Dermatology Life Quality Index(DLQI). DLQI is the widely used tool for the measurement of skin-health-related quality of life. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions in over 80 countries and is available in over 90 languages.This is a scale of how bad a person's skin disease affecting his/her life. The scale ranges from 0 (best) -10 (worst).
The effect of metformin on glucose and insulin metabolism as assessed by serum marker, HOMA index | baseline, Week 12
  HOMA index is calculated from serum glucose and insulin. The marker of glucose and insulin metabolism will be reported with pre- and post-metformin values compared.
Number of Participants Achieving a Greater Than or Equal to 90 Percentage Improvement From Baseline in Psoriasis Area and Severity Index (PASI 90) Score at Week 12 | baseline, Week 12
  Number of participants achieving greater than or equal to 90 percentage improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12. PASI is the widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) -72 (worst).
The effect of metformin on glucose and insulin metabolism as assessed by clinical marker, weight (kg) | baseline, Week 12
  The clinical marker will be reported with pre- and post-metformin values compared.
The effect of metformin on gut-microbiota profile of pre- and post-metformin samples | baseline, Week 12
  fecal macrobiotic profile.
  Comparison of gut microbiota in pre-and post-metformin samples.

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol; Statistical Analysis Plan (SAP); Informed Consent Form (ICF); Clinical Study Report (CSR) can be shared for the purpose of academic communication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Since the official start of the trial to the end of the trial
Access Criteria: Describe clearly about the reason of review.

REFERENCES:
- [Background] Wang X, Li R, Zhao X, Yu X, Sun Q. Metformin Promotes HaCaT Cell Apoptosis through Generation of Reactive Oxygen Species via Raf-1-ERK1/2-Nrf2 Inactivation. Inflammation. 2018 Jun;41(3):948-958. doi: 10.1007/s10753-018-0749-z. PMID 29549478
- [Background] Singh S, Bhansali A. Randomized Placebo Control Study of Metformin in Psoriasis Patients with Metabolic Syndrome (Systemic Treatment Cohort). Indian J Endocrinol Metab. 2017 Jul-Aug;21(4):581-587. doi: 10.4103/ijem.IJEM_46_17. PMID 28670544
- [Background] Ip W, Kirchhof MG. Glycemic Control in the Treatment of Psoriasis. Dermatology. 2017;233(1):23-29. doi: 10.1159/000472149. Epub 2017 May 25. PMID 28538228
- [Background] Wu CY, Shieh JJ, Shen JL, Liu YY, Chang YT, Chen YJ. Association between antidiabetic drugs and psoriasis risk in diabetic patients: results from a nationwide nested case-control study in Taiwan. J Am Acad Dermatol. 2015 Jan;72(1):123-30. doi: 10.1016/j.jaad.2014.08.042. Epub 2014 Oct 16. PMID 25443628
- [Background] Badr D, Kurban M, Abbas O. Metformin in dermatology: an overview. J Eur Acad Dermatol Venereol. 2013 Nov;27(11):1329-35. doi: 10.1111/jdv.12116. Epub 2013 Feb 26. PMID 23437788
- [Background] Brauchli YB, Jick SS, Curtin F, Meier CR. Association between use of thiazolidinediones or other oral antidiabetics and psoriasis: A population based case-control study. J Am Acad Dermatol. 2008 Mar;58(3):421-9. doi: 10.1016/j.jaad.2007.11.023. Epub 2008 Jan 14. PMID 18194825
- [Background] Tan L, Zhao S, Zhu W, Wu L, Li J, Shen M, Lei L, Chen X, Peng C. The Akkermansia muciniphila is a gut microbiota signature in psoriasis. Exp Dermatol. 2018 Feb;27(2):144-149. doi: 10.1111/exd.13463. PMID 29130553
- [Background] Shin NR, Lee JC, Lee HY, Kim MS, Whon TW, Lee MS, Bae JW. An increase in the Akkermansia spp. population induced by metformin treatment improves glucose homeostasis in diet-induced obese mice. Gut. 2014 May;63(5):727-35. doi: 10.1136/gutjnl-2012-303839. Epub 2013 Jun 26. PMID 23804561